CLINICAL TRIAL: NCT02630732
Title: Back School or Brain School for Patients Undergoing Surgery for Lumbar Radiculopathy? A Randomized Controlled Trial With Two-year Follow-up
Brief Title: Back School or Brain School for Patients Undergoing Surgery for Lumbar Radiculopathy?
Acronym: B²asic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: B²asic1
Record Dates: First submitted 2015-11-25; First posted 2015-12-15 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Lumbar Radiculopathy
Keywords: Back School; Brain School; Lumbar surgery; Education
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brain School (Active Comparator): Pain Neuroscience Education Program
  Interventions: Behavioral: Brain school
- Back School (Active Comparator): Classical Back School
  Interventions: Behavioral: Back school

INTERVENTIONS:
Behavioral: Brain school — 2 sessions of education provided by a therapist. The first session one day before surgery, the other two days after surgery. Education contains physiology of the central nerve system and the pain system. Information about acute pain, chronic pain and central sensitisation.
  Other Names: pain education, perioperative pain neuroscience education
  Arms: Brain School
Behavioral: Back school — Two education sessions ( one day before surgery and two days after surgery) with information about the biomechanics of the lumbar spine, physiology of the spine and ergonomics.
  Other Names: classical back school
  Arms: Back School

SUMMARY:
The primary scientific objective of the study entails examining whether perioperative pain neuroscience education (PPNE or 'brain school') is more effective than classical back school in reducing pain and improving pain inhibition in patients undergoing surgery for spinal radiculopathy. A secondary objective implies examining whether PPNE is more effective than classical back school in imparting a behavioural change (i.e. decreasing postoperative healthcare expenditure for lumbar radiculopathy), improving functioning in daily life and improving surgical experience (=better prepared for surgery, surgery meeting their expectations) in patients undergoing surgery for spinal radiculopathy.

DETAILED DESCRIPTION:
Prior to this study on lumbar radiculopathy patients, the proposed CPM protocol with EEG recordings will be pre-tested on a group of twenty healthy subjects, who will be fully informed about the study and subsequently gave their consent to participate. The proof of concept is set up to evaluate the effectiveness of the protocol, more specifically the appearance of nociceptive evoked potentials induced by electrical stimulation and the load on the subjects, as well as the safety of the protocol.

Low back pain is a frequently reported problem in our community. In the absence of successful outcomes following conservative intervention, surgery (including lumbar discectomy) is a recommended, evidence-based treatment for lumbar radiculopathy. To prevent chronicity following spinal surgery, preoperative education seems to be warranted. Current preoperative education programs in the orthopaedic and neurosurgical domain typically rely on the biomedical model, including education about (spinal) anatomy and biomechanics (like done in 'back schools'), as well as detailing the surgical procedure. Preoperative education focussing on the biomedical model is ineffective, and can increase anxiety and fear of patients undergoing spinal surgery. Therefore, there is a need to reconsider the content of education provided to patients undergoing spinal surgery.

Patient recruitment. All patients scheduled for surgery for lumbar radiculopathy in the UZ Brussel will be invited to participate. Lumbar radiculopathy is defined as pain due to lumbosacral nerve root compression. The NICE guidelines describe this as unilateral leg pain worse than the current back pain. This pain radiates to the foot or toes, and goes together with numbness and paraesthesia in the same distribution, which is associated with motor neurological deficit. Patients undergoing surgery for lumbar radiculopathy (n ≥ 100), willing to participate (including willingness to comply with the predetermined follow-ups), are recruited.

Randomization and concealment Randomization will be done by a computer-generated randomization list. A list with patient numbers and the group allocation that results from this randomization procedure will be stored in a sealed envelope. All the assessments will be performed by the same two investigators.

Intervention. At least 50 patients undergoing surgery for lumbar radiculopathy should get the experimental treatment, i.e. perioperative pain neuroscience education (PPNE). All patients will receive usual care plus surgery for lumbar radiculopathy. PPNE will comprise of two treatment sessions delivered by one physiotherapist (verbal one-on-one) and an educational booklet. The first treatment session will be in the week before surgery, the second on day 2 following surgery. Each treatment session will last approximately 60 minutes.

Patients will receive pain neuroscience education and will have extensive possibilities to ask questions during the sessions. At the end of the first educational session, patients will receive the educational booklet about the neurophysiology of pain and will be asked to read it carefully once before and once following surgery. In addition, they will be asked to complete the interactive part in the book before the second session. The second educational session (postoperative) is highly individually-tailored as it will readdress the patient's illness perceptions, answers questions and discuss the way of applying the knowledge into the patient's daily life. Immediately after the second educational session the participants will be asked to complete the Neurophysiology of Pain Test.

Control intervention. At least 50 patients should undergo the control treatment. As is the case with patients from the experimental group, patients in the control group will receive usual care plus surgery for lumbar radiculopathy. In addition to this standard treatment received by all patients included in the study, they will receive back school. The amount of therapist-patient contact, the number of treatment sessions as well as the mode of administration will be identical in both treatment groups. The procedure of the control treatment is identical to the experimental treatment, apart from the content of the treatment, which is based on the clinical guidelines and several studies. The education covers the normal course of back pain.

Data collection. All assessments will be performed in the UZ Brussel. Baseline assessments will take place during the week prior to the surgery. Immediate treatment effects will be assessed at post-operative day 3. Short-term and intermediate follow-up assessments will take place at, respectively, 6 weeks and 6 months post-surgery. Twelve and 24 months after the surgery the long-term follow-up treatment effects will be investigated.

Statistical analysis. At baseline, correlation analyses will be performed in order to examine possible associations between preoperative endogenous analgesia and the psychological factors.

All postoperative data analyses will be based on the Intention-to-Treat principle (i.e. the baseline observation carried forward method). AN(C)OVA repeated measures analyses will be used to evaluate and compare treatment effects. Baseline data of the outcome measure of interest, age and gender will serve as covariates. Statistical, as well as clinical significant differences will be defined and the effect size will be determined. In addition, numbers needed to treat will be calculated. Again, correlation analyses will be performed to evaluate whether changes in any of the outcome measures are related to changes in the psychological factors.

ELIGIBILITY:
Inclusion Criteria:

* Surgery for radiculopathy
* Speaking and reading Dutch fluently
* 18-65 years old
* Continuing usual care ( no new treatment) 6 weeks preceding surgery and during trial

Exclusion Criteria:

* Surgery for another condition than radiculopathy
* Symptoms of cord compression
* Rheumatoid, endocrinological, neurological or psychiatric disorder
* Chronic illness characterized by chronic pain that is not under control
* New treatments 6 weeks preceding surgery
* Pregnancy (preceding year)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Self-reported pain assessed by the Visual Analogue Scale | Change between baseline(1 week before surgery) and 3 days post-surgery, baseline and 6weeks post-surgery, baseline to 6 months post-surgery, baseline to 12 months post-surgery and baseline to 24 months post-surgery
  Patients fill in the Visual Analogue Scale ( 0 no pain - 10 unbearable pain) for their perceived back and leg pain.
Electrical pain threshold measured with an constant current electrical stimulator (DS7A Digitimer) | Change between baseline(1 week before surgery) and 3 days post-surgery, baseline and 6weeks post-surgery, baseline to 6 months post-surgery, baseline to 12 months post-surgery and baseline to 24 months post-surgery
  Determination of the electrical pain threshold with an electrical stimulator at the Median Nerve and Sural Nerves of each patient.
Endogenous pain inhibition assessed by the conditioned pain modulation paradigm | Change between baseline(1 week before surgery) and 3 days post-surgery, baseline and 6weeks post-surgery, baseline to 6 months post-surgery, baseline to 12 months post-surgery and baseline to 24 months post-surgery
  Conditioned pain modulation will be tested with the electrical stimulator as test stimulus and the cold pressor (12 °C) as conditioning stimulus. The difference between the electrical pain threshold (baseline) and the electrical pain threshold during the cold pressor (baseline + cold pressor) is called the conditioned pain modulation effect.
Quantitative Electroencephalography (QEEG) for brain mapping | Change between baseline(1 week before surgery) and 3 days post-surgery, baseline and 6weeks post-surgery, baseline to 6 months post-surgery, baseline to 12 months post-surgery and baseline to 24 months post-surgery
  During the conditioned pain modulation a QEEG is administered to examine the differences in brain activation on the brain map between the time frames.

SECONDARY OUTCOMES:
Postoperative healthcare expenditure for lumbar radiculopathy will be investigated by consultation of medical notes. | The difference between 3 days post-surgery, 6weeks post-surgery, 6 months, 12 months and 24 months
  Postoperative healthcare expenditure includes the number of days spent in hospital following surgery and medical tests related to post-operative surgery.
Functional status and well-being with the Short Form Health Survey-36 items | 1 week before surgery (except for surgical experience), 3 days after surgery, 6weeks post operative, 6 months, 12 months and 24 months
Surgical experience assessed with statements about patients their spinal surgery/education experience with a level of agreement on a numerical scale from 1 "minimal" to 10 "maximal agreement". | The difference between 3 days post-surgery, 6weeks post-surgery, 6 months, 12 months and 24 months
  Surgical experience addresses the way the patient feels to be prepared for surgery, and the extent the surgery met patient's expectations.
Pain catastrophizing with the Dutch translation of the Pain Catastrophizing Scale | 1 week before surgery (except for surgical experience), 3 days after surgery, 6weeks post operative, 6 months, 12 months and 24 months
  The pain catastrophizing scale consists of 13 items describing different thoughts and feelings that individuals may experience when they are experiencing pain.
Pain hypervigilance with the Dutch Pain Vigilance and Awareness Questionnaire. | 1 week before surgery (except for surgical experience), 3 days after surgery, 6weeks post operative, 6 months, 12 months and 24 months
  The Pain Vigilance and Awareness Questionnaire is a 16-item measure of attention to pain that assesses awareness, consciousness, vigilance, and observation of pain.
Kinesiophobia with the Tampa Scale for Kinesiophobia | 1 week before surgery (except for surgical experience), 3 days after surgery, 6weeks post operative, 6 months, 12 months and 24 months
Socio-economic factors with a demographic questionnaire concerning their return to work, professional occupation, incomes and grade of education. | 1 week before surgery (except for surgical experience), 3 days after surgery, 6weeks post operative, 6 months, 12 months and 24 months
  Patients will be asked to fulfil a demographic questionnaire concerning their grade of education, professional occupation, incomes and return to work.
Self-reported healthcare expenditure for which diaries will be used. | The difference between 3 days post-surgery, 6weeks post-surgery, 6 months, 12 months and 24 months
  Self-reported healthcare expenditure includes the number of postsurgical treatments (e.g. pain killers, physiotherapy, psychotherapy, osteopathy).

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - Sint-Maarten, Duffel, Antwerpen
  - AZ Sint-Dimpna, Geel, Antwerpen
  - Universitair Ziekenhuis Brussel, Jette, Brussels Capital

REFERENCES:
- [Background] Butler D, Moseley GL. Explain pain: Adelaide: NOI Group Publishing; 2003.
- [Background] van Wilgen CP, Nijs J. Pijneducatie: een praktische handleiding voor (para)medici: Bohn Stafleu van Loghum; 2010.
- [Background] Louw A. Your Nerves Are Having Back Surgery. International Spine and Pain Institute, Minneapolis, U.S.A.; 2012.
- [Background] Louw A, Butler DS, Diener I, Puentedura EJ. Development of a preoperative neuroscience educational program for patients with lumbar radiculopathy. Am J Phys Med Rehabil. 2013 May;92(5):446-52. doi: 10.1097/PHM.0b013e3182876aa4. PMID 23478459
- [Background] Dolphens M, Nijs J, Cagnie B, Meeus M, Roussel N, Kregel J, Malfliet A, Vanderstraeten G, Danneels L. Efficacy of a modern neuroscience approach versus usual care evidence-based physiotherapy on pain, disability and brain characteristics in chronic spinal pain patients: protocol of a randomized clinical trial. BMC Musculoskelet Disord. 2014 May 8;15:149. doi: 10.1186/1471-2474-15-149. PMID 24885889
- [Background] Louw A LQ, Crous LCC. Preoperative education for lumbar surgery for radiculopathy. S Afr J Physiother. 2009;65:3 - 8.
- [Background] Kreiner DS, Hwang SW, Easa JE, Resnick DK, Baisden JL, Bess S, Cho CH, DePalma MJ, Dougherty P 2nd, Fernand R, Ghiselli G, Hanna AS, Lamer T, Lisi AJ, Mazanec DJ, Meagher RJ, Nucci RC, Patel RD, Sembrano JN, Sharma AK, Summers JT, Taleghani CK, Tontz WL Jr, Toton JF; North American Spine Society. An evidence-based clinical guideline for the diagnosis and treatment of lumbar disc herniation with radiculopathy. Spine J. 2014 Jan;14(1):180-91. doi: 10.1016/j.spinee.2013.08.003. Epub 2013 Nov 14. PMID 24239490
- [Background] Louw A, Diener I, Landers MR, Puentedura EJ. Preoperative pain neuroscience education for lumbar radiculopathy: a multicenter randomized controlled trial with 1-year follow-up. Spine (Phila Pa 1976). 2014 Aug 15;39(18):1449-57. doi: 10.1097/BRS.0000000000000444. PMID 24875964
- [Derived] Van Bogaert W, Huysmans E, Coppieters I, Nijs J, Putman K, Ickmans K, Moens M, Goudman L, Stas L, Buyl R. The Mediating Role of Pain Cognitions and Pain Sensitivity in the Treatment Effect of Perioperative Pain Neuroscience Education in People Undergoing Surgery for Lumbar Radiculopathy. J Pain. 2024 Aug;25(8):104521. doi: 10.1016/j.jpain.2024.03.017. Epub 2024 Apr 2. PMID 38575104
- [Derived] Van Bogaert W, Coppieters I, Nijs J, Buyl R, Ickmans K, Moens M, Goudman L, Putman K, Huysmans E. Influence of Preoperative Pain, Cognitions, and Quantitative Sensory Testing Measures on the Effects of Perioperative Pain Neuroscience Education for People Receiving Surgery for Lumbar Radiculopathy: Secondary Analysis of a Randomized Controlled Trial. J Orthop Sports Phys Ther. 2024 Apr;54(4):279-288. doi: 10.2519/jospt.2024.12051. PMID 38189683
- [Derived] Huysmans E, Goudman L, Coppieters I, Van Bogaert W, Moens M, Buyl R, Nijs J, Louw A, Logghe T, Putman K, Ickmans K. Effect of perioperative pain neuroscience education in people undergoing surgery for lumbar radiculopathy: a multicentre randomised controlled trial. Br J Anaesth. 2023 Sep;131(3):572-585. doi: 10.1016/j.bja.2023.05.007. Epub 2023 Jun 19. PMID 37344337
- [Derived] Van Bogaert W, Putman K, Coppieters I, Goudman L, Nijs J, Moens M, Buyl R, Ickmans K, Huysmans E. Health-related quality of life deviations from population norms in patients with lumbar radiculopathy: associations with pain, pain cognitions, and endogenous nociceptive modulation. Qual Life Res. 2022 Mar;31(3):745-757. doi: 10.1007/s11136-021-02964-5. Epub 2021 Aug 3. PMID 34342846